CLINICAL TRIAL: NCT01329991
Title: A Phase 1b Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Drug-Drug Interaction of PLX5622 in Patients With Rheumatoid Arthritis Who Are Receiving Methotrexate
Brief Title: Phase 1b Study of PLX5622 in Rheumatoid Arthritis Patients Who Are Receiving Methotrexate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plexxikon (Industry)
Responsible Party: Keith Nolop, MD, Plexxikon
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLX115-02
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PLX5622

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- oral dose of 200 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take an oral dose of PLX5622 for 14 days and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- oral dose of 400 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take an oral dose of PLX5622 for 14 days and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- oral dose of 800 mg PLX5622 (Active Comparator): 6 subjects will be randomized to take an oral dose of PLX5622 for 14 days and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- oral dose of PLX5622-dose to be determined (Active Comparator): 6 subjects will be randomized to take an oral dose of PLX5622 for 14 days and 2 subjects will be randomized to take placebo.
  Interventions: Drug: PLX5622
- Placebo Comparator (Placebo Comparator): 2 patients per cohort will be randomly assigned to take placebo. 8 patients total will be randomized to take placebo in this study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLX5622 — PLX5622 drug substance is an achiral,small molecule Fms kinase inhibitor. The drug product is available in capsule form, to be taken orally, in a dosage strength of 100 mg with matching placebo
  Arms: oral dose of 200 mg PLX5622; oral dose of 400 mg PLX5622; oral dose of 800 mg PLX5622; oral dose of PLX5622-dose to be determined
Drug: Placebo — Matching placebo for PLX5622
  Arms: Placebo Comparator

SUMMARY:
PLX115-02 is a phase 1b study to assess how the study drug, PLX5622: 1. affects the body, 2. how the body affects PLX5622 3. the interaction of PLX5622 with Methotrexate and 4. the safety of PLX5622 in rheumatoid arthritis patients taking Methotrexate

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years old with a diagnosis of rheumatoid arthritis by ACR criteria for ≥ 3 months.
* Prior to Day 1, patients must be on oral or subcutaneous methotrexate (≥10 mg/week and ≤ 25 mg/week) for at least 12 weeks (with a stable dose for at least 4 weeks) and folate (≥ 5 mg/week) for at least 6 weeks, and willing to continue on this regimen for the duration of the study.
* Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥ 1.5 X 109/L, Hgb > 9 g/dL, platelet count ≥ 100 X 109/L, AST/ALT WNL, albumin ≥ 3 g/dL, calculated CrCl>60 mL/min using Cockcroft-Gault formula).
* Women of child-bearing potential must have a negative pregnancy test within 7 days prior to initiation of dosing with study drug and must agree to use a double barrier method of birth control from the time of the negative pregnancy test up to 30 days after the last dose of study drug. Women of nonchildbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year.
* Fertile men must agree to use an acceptable method of birth control while on study drug. Acceptable methods of contraception must include either abstinence from the first dose of study drug through 4 weeks after the last dose of study drug, or use of a condom with instructions to the female partner of child-bearing potential to also be protected as above.
* Willing and able to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

* Use of biologic response modifiers within the following periods prior to Day 1: 4 weeks for Kineret (anakinra) and Enbrel (etanercept); 12 weeks for Remicade (infliximab), Humira (adalimumab), Simponi (golimumab), Orencia (abatacept), Actemra (tocilizumab), or Cimzia (certolizumab); 12 months for Rituxan (rituximab).
* Use of Arava (leflunomide) within 12 weeks prior to Day 1 or any immunosuppressive agents, including hydroxychloroquine or sulfasalazine, within 4 weeks of Day 1.
* Investigational drug use within 4 weeks of Day 1.
* Positive urine drug screen for drugs of abuse (except for opiates if being used for RA).
* Concomitant use of DMARDs (other than methotrexate), biological response modifiers, or known strong inducers or inhibitors of CYP3A4 (see Appendix 2).
* Uncontrolled intercurrent illness.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* QTc ≥ 450 msec at Screening.
* The presence of a medical or psychiatric condition that, in the opinion of the Principal Investigator, makes the patient inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety-Number of patients with adverse events | 22 days
  Subjects will take oral doses of PLX5622 once a day for 14 days. Physical examinations, vital signs, 12-lead electrocardiograms (ECG), adverse events, hematology, serum chemistry, coagulation, and urinalysis will be used to assess safety throughout Day 1-14 of the study, Day 17 and the follow up study visit on day 22. Adverse events will be monitored and reviewed for safety issues/abnormal changes in the above mentioned tests.

SECONDARY OUTCOMES:
Pharmacokinetic profile: Measurement of area under the plasma-concentration-time curve | 22 days
  The pharmacokinetic profile of plasma PLX5622 and Methotrexate will be analyzed by measurement of area under the plasma concentration-time curve [AUC0-t, AUC0-inf, AUC0-24].
Pharmacokinetic evaluation: Measurement of Peak Concentration | 22 days
  The pharmacokinetic profile of plasma PLX5622 and Methotrexate will be analyzed by measurement of peak concentration (Cmax) and time to peak concentration (Tmax).
Pharmacokinetic profile: Measurement of half life, apparent systemic clearance, and apparent volume of distribution, terminal phase. | 22 days
  The pharmacokinetic profile of plasma PLX5622 and Methotrexate will be analyzed by measurement of half-life (T1/2), apparent systemic clearance (CL/F), and apparent volume of distribution, terminal phase (Vz/F).
Pharmacodynamics-Effect of PLX5622 on the body | 22 days
  The effects of PLX5622 on the body will be measured by observing early response biomarkes of disease activity.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pinnacle Research Group, Anniston, Alabama
  - Medical Practice of Justus Fiechtner, MD, Lansing, Michigan
  - Altoona Center for Clinical research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas